CLINICAL TRIAL: NCT00557336
Title: Evaluation of Efficacy and Safety of Somatropin in SGA Children Due to IUGR
Brief Title: Efficacy and Safety of Growth Hormone Treatment in Children Small for Gestational Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHLIQUID-1523
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Foetal Growth Problem; Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to evaluate the height gain during 12 months of growth hormone treatment in children born small for gestational age due to intrauterine growth retardation.

ELIGIBILITY:
Inclusion Criteria:

* Born small for gestational age (SGA) due to intrauterine growth retardation (IUGR) defined as birth length and/or weight below P10
* Chronological age at least 4 years old until bone age maturation of maximum 12 years for girls and maximum 13,5 for boys at time of inclusion in the study
* Insufficient catch-up growth (height lesser than or equal to -2.5 SDS for chronological age
* Normal response to GH stimulation test (greater than 10 ng/mL)

Exclusion Criteria:

* Diabetes
* Growth retardation associated with infections severe chronic diseases (including chromosomal anomaly or nutritional disorders)
* Treatment with any medical product (anabolic drugs, sex steroids, etc.) which may interfere with GH effects
* History or presence of severe disease that could interfere with GH treatment/participation in the trial, e.g. active malignancy
* Previous or ongoing growth hormone therapy

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2003-07-28 (Actual); Primary Completion 2005-06-29 (Actual); Study Completion 2005-06-29 (Actual)

PRIMARY OUTCOMES:
Height gain according to birth group, age of onset, the treatment and Tanner stage | during 12 months of treatment

SECONDARY OUTCOMES:
Height SDS for bone age | during 12 months of treatment
Height velocity SDS for bone age | during 12 months of treatment
Height velocity for chronological age | during 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (33):
- Spain (33):
  - Novo Nordisk Investigational Site, Albacete
  - Novo Nordisk Investigational Site, Alicante
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Badajoz
  - Novo Nordisk Investigational Site, Badalona
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Calella de La Costa
  - Novo Nordisk Investigational Site, Cáceres
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, El Palmar
  - Novo Nordisk Investigational Site, Elche
  - Novo Nordisk Investigational Site, Esplugues Llobregat
  - Novo Nordisk Investigational Site, Getafe
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Granollers
  - Novo Nordisk Investigational Site, Huelva
  - Novo Nordisk Investigational Site, Jaén
  - Novo Nordisk Investigational Site, Las Palmas
  - Novo Nordisk Investigational Site, Leganés
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Martorell
  - Novo Nordisk Investigational Site, Mataró
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Pamplona
  - Novo Nordisk Investigational Site, Sabadell
  - Novo Nordisk Investigational Site, Salamanca
  - Novo Nordisk Investigational Site, Santa Cruz de Tenerife
  - Novo Nordisk Investigational Site, Santander
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Tarrasa
  - Novo Nordisk Investigational Site, Vitoria-Gasteiz
  - Novo Nordisk Investigational Site, Zaragoza

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com